CLINICAL TRIAL: NCT03649152
Title: A Phase 2a, Double-Blind, Randomized, Placebo-Controlled, Crossover Study Evaluating the Safety and Efficacy of Propagermanium in Patients With Primary Focal Segmental Glomerulosclerosis (FSGS) Who Are Receiving Irbesartan
Brief Title: Safety and Effectiveness of Propagermanium in Focal Segmental Glomerulosclerosis Participants Receiving Irbesartan
Acronym: ACTION
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dimerix Bioscience Pty Ltd (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DMX-200-202 A; ACTRN12618000910202p (Registry Identifier: Australia New Zealand Clinical Trials Registry)
Record Dates: First submitted 2018-08-07; First posted 2018-08-28 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2020-02

CONDITIONS: Focal Segmental Glomerulosclerosis
MeSH Terms: conditions — Glomerulosclerosis, Focal Segmental | interventions — propagermanium

STUDY DESIGN:
Intervention Model Description: Double-blind, Randomised, Placebo-Controlled, Crossover Study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propagermanium then Placebo (Experimental): Propagermanium one capsule orally twice daily for 16 weeks. Compliance will be measured by drug accountability and completion of a participant diary.
  Participants will receive 16 weeks propagermanium and 16 weeks placebo separated by a 6 week washout period.
  Interventions: Drug: Propagermanium; Drug: Placebo
- Placebo then Propagermanium (Experimental): Propagermanium one capsule orally twice daily for 16 weeks. Compliance will be measured by drug accountability and completion of a participant diary.
  Participants will receive 16 weeks placebo and 16 weeks propagermanium separated by a 6 week washout period.
  Interventions: Drug: Propagermanium; Drug: Placebo

INTERVENTIONS:
Drug: Propagermanium — Immediate release capsule
  Other Names: PPG; repagermanium; DMX-200
Drug: Placebo — Placebo capsule

SUMMARY:
This study will be evaluating the safety and efficacy of propagermanium for the treatment of participants with FSGS who are already taking irbesartan by:

* monitoring symptoms that participants may experience while on the study,
* measuring levels of protein in participant's urine and kidney function during the course of the study,
* measuring the levels of propagermanium and irbesartan that enters into participant's urine and blood, and
* comparing the propagermanium outcomes to participants' pre-study and placebo outcomes.

Eligible participants will randomly be assigned to one of two arms to receive both the propagermanium and placebo in different orders as follows, either:

Treatment Period 1 taking a propagermanium capsule twice a day for 16 weeks, followed by a six week washout period followed by Treatment Period 2 taking a placebo capsule twice a day for 16 weeks.

OR Treatment Period 1 taking a placebo capsule twice a day for 16 weeks, followed by a six week washout period followed by Treatment Period 2 taking a propagermanium capsule twice a day for 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 80 (inclusive) at screening;
2. A diagnosis of primary FSGS confirmed by renal biopsy;
3. Must be receiving a stable dose of 300 mg daily dose of irbesartan (in any marketed formulation) for at least 3 months prior to screening, and have no plan to change treatment regime throughout the study;
4. Patients can be on stable doses of angiotensin converting enzyme inhibitors, aldosterone inhibitors, direct renin inhibitor and/or sodium-glucose co-transporter- 2 inhibitors. However, the dose and regimen must be stable for 3 months prior to screening and must have no plan to change treatment regime throughout the study.
5. If taking immunosuppressive medications (except for rituximab or cyclophosphamide), must have a stable treatment regime for 3 months prior to screening and do not have plans to alter the regimen except to maintain therapeutic immunosuppression or in the event of adverse events. Patients who have received rituximab or cyclophosphamide must have ceased treatment for at least 6 months prior to screening;
6. Mean of two protein/creatinine ratio values (screening and baseline) of ≥ 1326 mg/g (150 mg/mmol), and within ± 30% of the screening value at the baseline assessment;
7. Estimated glomerular filtration rate ≥ 25 mL/min/1.73 m^2 using chronic kidney disease epidemiology collaboration (CKD-EPI) formula at screening;
8. Serum potassium levels (screening and baseline) < 5.5 mmol/L. If either value is 5.5 or above, the patient may receive dietary advice and be retested 1 week later;
9. A female patient is eligible to participate if she is not pregnant, not breastfeeding, and at least 1 of the following conditions applies:

   * Not of childbearing potential, defined as surgically sterile (documented hysterectomy, bilateral salpingectomy or bilateral oophorectomy) or postmenopausal (no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone [FSH] level in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy; however, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient.);
   * Of childbearing potential and agrees to use a highly effective method of contraception consistently during the treatment period and for at least 60 days after the last dose of investigational product;
10. A male patient with a female partner of childbearing potential is eligible to participate if he agrees to use acceptable contraception during the treatment period and for at least 60 days after the last dose of investigational product and refrains from donating sperm during this period;
11. Have given written informed consent prior to any study procedures being performed.

Exclusion Criteria:

1. Has FSGS secondary to another condition;
2. A history of type 1 diabetes mellitus, diagnosis of type 2 diabetes mellitus prior to FSGS positive renal biopsy, or non-fasting blood glucose > 180 mg/dL (10 mmol/L) at screening;
3. A prior kidney organ or stem cell transplant;
4. A major adverse cardiac event within 6 months before screening;
5. Lymphoma, leukaemia, or any malignancy within the past 5 years except for basal cell or squamous cell carcinomas of the skin or cervical carcinoma in situ that have been resected with no evidence of metastatic disease for 3 years;
6. Jaundice, active hepatitis, or known hepatobiliary disease (except asymptomatic cholelithiasis);
7. Alanine aminotransferase and/or aspartate aminotransferase more than two times the upper limit of normal at screening;
8. Participation in any clinical study with an experimental medication or device within 90 days or 5 half-lives (whichever is longer) of screening or have previously participated in a study involving propagermanium;
9. Positive screening assessment for viral hepatitis B surface antigen or hepatitis C virus (HCV) antibody AND positive HCV RNA or human immunodeficiency virus (HIV), or a history of illicit drug injecting;
10. Seated blood pressure of ≥ 160/100 mmHg at screening;
11. Body mass index ≥ 35 kg/m^2 at screening;
12. Past hospitalisation for a major depressive episode;
13. Is breast feeding or pregnant;
14. Unable to comply with the study procedures and assessments, including the ability swallow capsules;
15. Any other disease, physical or psychological condition that the investigator or sponsor believes may contraindicate the use of the investigational medicinal product or affect the interpretation of study results or render the patient at high risk from treatment complications;
16. Are investigator site personnel directly affiliated with this study and their immediate families. Immediate family is defined as a spouse, parent, child or sibling, whether biological or legally adopted.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-11-08 (Actual); Primary Completion 2020-06-16 (Actual); Study Completion 2020-07-13 (Actual)

PRIMARY OUTCOMES:
The Number of Adverse Events with the Adjunct use of Propagermanium Compared to Placebo in Participants with FSGS who are Receiving Irbesartan | Sixteen weeks
  Assessed by monitoring of adverse events

SECONDARY OUTCOMES:
The Frequency of Proteinuria-Based Responses to Treatment Compared to Placebo | Sixteen weeks
  Assessed by testing a 24-hour urine sample.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Roger, MD, Principal Investigator — Renal Research
Locations (11):
- Australia (11):
  - Renal Research, Gosford, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Westmead, Westmead, New South Wales
  - Sunshine Coast University Hospital, Birtinya, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Box Hill Hospital, Box Hill, Victoria
  - Austion Hospital, Heidelberg, Victoria
  - Sunshine Hospital, Melbourne, Victoria
  - Melbourne Renal Research Group, Melbourne, Victoria
  - Epworth Hospital, Richmond, Victoria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hodson EM, Sinha A, Cooper TE. Interventions for focal segmental glomerulosclerosis in adults. Cochrane Database Syst Rev. 2022 Feb 28;2(2):CD003233. doi: 10.1002/14651858.CD003233.pub3. PMID 35224732